CLINICAL TRIAL: NCT05060315
Title: EVOLVE: a Virtual, Observational, Patient-Centric Prospective Study to Evaluate Real-World Use of Next Generation Infusion Pumps to Administer Remodulin to Patients with Pulmonary Arterial Hypertension
Brief Title: Evaluate Real-World Use of Next Generation Infusion Pumps to Administer Remodulin
Acronym: EVOLVE
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: REM-PH-417
Record Dates: First submitted 2021-04-06; First posted 2021-09-29 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- De Novo Cohort: Patients new to parenteral prostacyclin-class therapy.
  Interventions: Combination Product: Remunity Pump for Remodulin
- Transition Cohort: Patients who had been receiving SC treprostinil therapy via a previous generation infusion pump prior to transitioning to a next generation infusion pump.
  Interventions: Combination Product: Remunity Pump for Remodulin

INTERVENTIONS:
Combination Product: Remunity Pump for Remodulin — Participants on the study will receive Remodulin via the Remunity Pump with dosing and titration managed at the discretion of the prescribing healthcare professional. Dosing and titration of Remodulin will in no way be influenced by the participation in this study or this protocol.

SUMMARY:
To observe and assess drug administration activities, time spent on drug administration activities, and patient-reported outcomes (PROs) including quality of life, treatment satisfaction, and patient perception of devices related to use of United Therapeutics Corporation (UTC)-developed next-generation infusion pumps to administer Remodulin in patients with Pulmonary Arterial Hypertension (PAH).

DETAILED DESCRIPTION:
This is a virtual, patient-centric, observational study that will follow approximately 60 participants through 8 weeks following initiation of Remodulin therapy via their UTC-developed next generation infusion pump and consists of remote and electronic assessments administered to patient via the uMotif® data capture platform at Study Enrollment, Week 2, Week 4, and Week 8 or Early Withdrawal (if applicable).

The study population will consist of 2 cohorts of PAH patients:

1. De Novo Cohort: patients new to parenteral prostacyclin-class therapy.
2. Transition Cohort: patients who had been receiving SC treprostinil therapy via a previous generation infusion pump prior to transitioning to a next generation infusion pump.

The De Novo Cohort will initiate subcutaneous (SC) Remodulin via a next generation infusion pump as prescribed by their healthcare professional. Participants will be followed from day of Study Enrollment, which will be Day 1, through 8 weeks while using next generation infusion pump, or until discontinuation of Remodulin (early withdrawal), whichever comes first.

The Transition Cohort will have previously been receiving SC treprostinil utilizing a previous generation infusion pump prior to transitioning to delivery of Remodulin via next generation infusion pump, as prescribed by their healthcare provider. Participants will be followed from day of Study Enrollment, which will be Day 1, through 8 weeks while using next generation infusion pump, or until discontinuation of Remodulin (early withdrawal), whichever comes first.

Following the completion of study assessments at Week 8 or Early Withdrawal (if applicable), participants will continue Remodulin therapy via their infusion pump at their prescriber's discretion.

ELIGIBILITY:
Inclusion Criteria - De Novo Cohort:

1. The patient is greater than 22 years of age at time of providing informed consent.
2. The patient is willing and able to provide informed consent and has the ability to answer surveys, questionnaires, and use the diary in English.
3. The patient has started SC Remodulin via the Remunity Pump for Remodulin (treprostinil) Injection prior to providing informed consent.
4. The patient has not been previously treated with a parenteral prostacyclin-class therapy in the past 30 days prior to initiating SC Remodulin therapy with the Remunity Pump, except in cases where the patient initiates inpatient parenteral prostacyclin-class therapy via another infusion pump and subsequently started SC Remodulin therapy with the Remunity Pump for Remodulin (treprostinil) Injection in the outpatient setting.

Inclusion Criteria - Transition Cohort:

1. The patient is greater than 22 years of age at time of providing informed consent.
2. The patient is willing and able to provide informed consent and has the ability to answer surveys, questionnaires, and use the diary in English.
3. The patient has started SC Remodulin via the Remunity Pump for Remodulin (treprostinil) Injection prior to providing informed consent.
4. The patient had been receiving continuous infusion of SC treprostinil via an infusion pump other than Remunity for at least 60 days prior to initiating SC Remodulin therapy with the Remunity Pump.

Exclusion Criteria:

1. The patient is pregnant, trying to become pregnant, or lactating.
2. For those in the Transition Cohort: The patient has a history of adverse events resulting from interruptions in their treprostinil infusions over relatively short periods (such as less than 8 hours) as they may be at higher risk in the event of pump failure, especially at night.
3. The patient is enrolled in, has participated within the last 30 days, or is planning to participate in an interventional study. Note: co-enrollment in other observational studies is permitted.
4. For those in the Transition Cohort: The patient had been receiving parenteral treprostinil via IV administration prior to transitioning to the Remunity Pump.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 60 participants in the United States will be enrolled in this study. Participants new to parenteral prostacyclin-class therapy prior to initiating next generation pump for Remodulin will be enrolled in the De Novo Cohort. Participants that had received SC treprostinil therapy via a previous generation infusion pump prior to transitioning to delivery of SC Remodulin via a next generation infusion pump will be enrolled in the Transition Cohort. The number of participants in each cohort will be assessed throughout the duration of study and may be refined accordingly.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To observe and assess time spent on drug administration activities related to the United Therapeutics Corp.-developed next generation pumps to administer Remodulin in patients with PAH | 8 Weeks
  Participants will be asked to participate in a comprehensive collection of the drug administration activities data consisting of a 7-day evaluation period of daily drug administration activities pertaining to their next generation infusion pump via the Drug Administration Activities Diary.
To observe and assess patient reported outcomes via the Pulmonary Hypertension Functional Class Self-Report | 8 Weeks
  Participant self-assessment of Functional Class (I to IV) will be performed using the Pulmonary Hypertension Functional Class Self-Report (PH-FC-SR), as adapted from the pulmonary hypertension World Health Organization Functional Classification System.
To observe and assess patient reported outcomes via the Patient Perception of Parenteral Infusion System Questionnaire | 8 Weeks
  The Patient Perception of Parenteral Infusion System Questionnaire will be administered to assess the participant's perception of their infusion pumps.
To observe and assess patient reported outcomes via the Abbreviated Treatment Satisfaction Questionnaire for Medication | 8 Weeks
  The Abbreviated Treatment Satisfaction Questionnaire for Medication (TSQM-9) is a validated instrument to assess participants' satisfaction with medication, providing scores on 3 scales - effectiveness, convenience, and global satisfaction.
To observe and assess patient reported outcomes via the emPHasis-10 questionnaire | 8 Weeks
  The emPHasis-10 questionnaire is a reliable and validated tool for assessment of health-related quality of life in pulmonary hypertension. It consists of 10 items, which address breathlessness, fatigue, control, and confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Morrisville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No